CLINICAL TRIAL: NCT07092566
Title: Efficacy of Ropivacaine Epinephrine Clonidine Ketorolac (R.E.C.K) vs Exparel in Robotic Nephrectomy: a Randomized, Prospective Trial
Brief Title: R.E.C.K vs Exparel in Robotic Nephrectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00133736; ONC-GU-2404 (Other: AHWFBCCC)
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Renal Carcinoma; Nephrectomy / Methods; Pain Management
Keywords: Analgesics; Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell; Agnosia | interventions — Ropivacaine; Epinephrine; Clonidine; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Intraoperative R.E.C.K.
  Interventions: Drug: Ropivacaine HCL; Drug: Epinephrine; Drug: Clonidine HCL; Drug: Ketorolac
- Arm B (Experimental): Intraoperative Exparel
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Ropivacaine HCL — 123 mg, intramuscular
  Arms: Arm A
Drug: Exparel — 100 mL total dose - Intramuscular (IM), intraoperatively
  Other Names: bupivacaine liposome injectable suspension
  Arms: Arm B
Drug: Epinephrine — 0.25 mg, intramuscular
  Arms: Arm A
Drug: Clonidine HCL — 0.04 mg, intramuscular
  Arms: Arm A
Drug: Ketorolac — 15 mg, intramuscular
  Arms: Arm A

SUMMARY:
The purpose of the study is to evaluate the efficacy of R.E.C.K (ropivacaine epinephrine clonidine ketorolac) vs Exparel during robotic partial and radical nephrectomy in a single institution, prospective, randomized trial. The study will evaluate post operative Numerical Rating Score (NRS) pain scores, post operative pain medication intake (opioids and over-the-counter pain medicines) and length of stay across the two patient cohorts. The findings will help to inform whether the increased cost of Exparel when compared to R.E.C.K is justified.

DETAILED DESCRIPTION:
Intra-op opioid administration will be collected and recorded for each participant via EMR review. While in the post anesthesia care unit and the remainder of the inpatient stay, the following will be assessed and captured: pain score via Numerical Rating Score (NRS) captured per standard of care, oral and IV opioid intake, and length of inpatient stay.

After discharge, the participants will be asked to record and timestamp the following in a provided take-home paper diary: pain via NRS in response to the prompt "How much pain are you experiencing right now?" and self-administered medications and dose (ibuprofen, acetaminophen, naproxen, and opioids) throughout the day.

Treatment will be administered intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an IRB-approved informed consent
2. Age ≥ 18 years at the time of consent.
3. Planned robotic partial or radical nephrectomy

Exclusion Criteria:

1. Determined not to be a candidate to receive R.E.C.K or Exparel per the enrolling investigator
2. Known pregnancy
3. Chronic opioid use within 30 days (as per patient report) prior to randomization (defined as ≥ 30 MME/day)
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator.
5. Known allergy to R.E.C.K. and/or Exparel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) pain intensity scores through 7 days (168 hours) for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 7 Post-Surgery
  Assess pain intensity (evaluated by NRS) after surgery on the as response to the prompt: "On a scale of 0 to 10, where 0 = no pain and 10 = worst possible pain, how much pain are you having right now?" The AUC will be derived for each participant from self-reported pain scores and will be summarized by treatment group. Generalized linear models with main effect of treatment will be estimated to test for significant differences in AUC between the arms.

SECONDARY OUTCOMES:
Estimated difference in Numeric Rating Scale (NRS) pain intensity scores over 7 days for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 7 Post-Surgery
  Assess modeled daily pain scores using repeated measures analysis; the primary comparison is the treatment-by-time interaction effect. The NRS is a scale to evaluate pain in response to the prompt "On a scale of 0 to 10, where 0 = no pain and 10 = worst possible pain, how much pain are you having right now?"
Total postsurgical opioid consumption (morphine equivalent dose) over 7 days for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 7 Post-Surgery
  Total opioid consumption will be calculated for each participant as the sum of all administered opioid doses from Postoperative Day 0 through Day 7. All opioid doses will be converted to morphine equivalent dose (MED) using standard conversion factors. The total MED will be compared between treatment arms .
Estimated difference in postsurgical opioid consumption (in morphine equivalent dose) over 7 days for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 7 Post-Surgery
  Assess modeled daily postsurgical opioid consumption using repeated measures analysis; the primary comparison is the treatment-by-time interaction effect. Daily totals in morphine equivalent dose will be calculated for each participant.
Total postsurgical non-opioid pain medication consumption (in milligrams) over 7 days for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 7 Post-Surgery
  Total milligrams consumed for each for ibuprofen, acetaminophen, and naproxen will be calculated for each participant as the sum of the total milligrams consumed from Post Operative Day 0 trough Post Operative Day 7 and compared between arms. The total milligrams consumed will be compared between treatment arms.
Estimated difference in postsurgical non-opioid consumption over 7 days for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 7 Post-Surgery
  Assess modeled daily postsurgical non-opioid consumption using repeated measures analysis; the primary comparison is the treatment-by-time interaction effect. Medications informing this analysis include ibuprofen, acetaminophen, and naproxen. Daily totals in milligrams consumed will be calculated for each participant.
Proportion of opioid-free participants after 7 days for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 7 Post-Surgery
  The proportion of participants who did not receive any opioid medication from Postoperative Day 0 through Day 7. Participants will be classified as opioid-free if their total opioid consumption during this period is zero (0 mg morphine equivalent dose). The proportion will be compared between treatment arms.
Time to first opioid intake in hours from surgery for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 7 Post-Surgery
  Time to first opioid intake will be defined as the time, in hours, from end of surgery to first opioid medication taken. If participant does not use opioid medication, the time to first opioid intake will be censored at the end of POD7. This will be compared between the arms.
Length of inpatient stay after surgery for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 30 Post-Surgery
  Length of inpatient stay is defined as the total duration, in days (where a full day includes an overnight stay), from the end of surgery until the participant is formally discharged from the hospital. This measure will be used to compare hospitalization duration between treatment arms.

OTHER OUTCOMES:
Proportion of participants experiencing any study -drug related adverse events within 30 days of surgery for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 30 Post-Surgery
  A binary variable indicating experience of at least one AE occurring within 30 days of administration of study drug will be determined for each participant. The proportions will be compared between treatment arms.
Proportion of participants experiencing any study -drug related Grade 3+ adverse events within 30 days of surgery for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 30 Post-Surgery
  A binary variable indicating experience of at least one Grade 3+ AE occurring within 30 days of administration of study drug will be determined for each participant. The proportions will be compared between treatment arms.
Proportion of participants experiencing any serious adverse events within 30 days of surgery for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 30 Post-Surgery
  A binary variable indicating experience of at least one SAE occurring within 30 days of administration of study drug will be determined for each participant. The proportions will be compared between treatment arms.
Proportion of participants experiencing any surgical complications within 14 days of surgery for participants receiving Exparel vs. R.E.C.K. | Day of Surgery to Day 14 Post-Surgery
  A binary variable indicating experience of at least one surgical complication occurring within 14 days of administration of study drug will be determined for each participant. The proportions will be compared between treatment arms.
Proportion of participants experiencing post-discharge readmission within 30 days of initial discharge for participants receiving Exparel vs. R.E.C.K. | Day of Discharge to Day 30 Post-Discharge
  A binary variable indicating post-discharge readmission within 30 days of initial hospital discharge will be determined for each participant. The proportions will be compared between treatment arms.
All-cause mortality within 30 days post-surgery for participants receiving Exparel vs. R.E.C.K. | Day of Discharge to Day 30 Post-Discharge
  The proportions of participants alive at 30 days after initial hospital discharge will be compared between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Ornob, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No